CLINICAL TRIAL: NCT07281586
Title: Step-down Therapy After Long-term Osteoporosis Treatment: A Randomized Trial
Brief Title: Step-down Therapy After Long-term Osteoporosis Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202412063MINE
Record Dates: First submitted 2025-11-25; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis
Keywords: long-term denosumab; zoledronate; half-dose denosumab; de-escalation strategy
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Zoledronate is given 6 months after the final denosumab injection, with a second zoledronate infusion administered 18 months after the last denosumab dose.
  Interventions: Drug: zoledronate
- Denosumab De-escalation + Zoledronate (Experimental): Half-dose denosumab plus zoledronic acid at 6 months after the last denosumab dose, followed by a second half-dose denosumab injection at 12 months and a second zoledronic acid infusion at 18 months after the final denosumab dose.
  Interventions: Drug: zoledronate; Drug: Denosumab De-escalation

INTERVENTIONS:
Drug: zoledronate — In the control arm, participants will receive zoledronate at trial entry, with a second dose administered at the start of the second year
  Arms: Control
Drug: zoledronate — In the intervention arm, participants will receive zoledronate at trial entry, with a second dose administered at the start of the second year.
  Arms: Denosumab De-escalation + Zoledronate
Drug: Denosumab De-escalation — In the intervention arm, participants will receive a half-dose of denosumab at trial entry, followed by a second half-dose 6 months later during the first year.
  Arms: Denosumab De-escalation + Zoledronate

SUMMARY:
Maintaining bone mineral density (BMD) after discontinuing denosumab (Prolia) is a major clinical challenge, as rapid bone loss commonly occurs when treatment is stopped, especially after more than three years of use. Standard sequential therapy with bisphosphonates such as zoledronic acid (Aclasta) often fails to fully prevent BMD decline, and most bone loss occurs within the first year, making effective suppression of the rebound effect essential.

This study investigates whether a de-escalation strategy-using half-dose denosumab (30 mg every six months) combined with sequential zoledronic acid-can better preserve lumbar spine BMD after long-term denosumab therapy. Eligible participants include postmenopausal women and men ≥50 years old with osteoporosis or osteopenia-related fractures who have received ≥3 years of denosumab.

The open-label trial applies stratified randomization based on denosumab duration (<4 years vs. ≥4 years), assigning 22 participants to each group.

Control group: standard therapy with one zoledronic acid infusion at the end of denosumab's effect and a second infusion one year later.

Intervention group: half-dose denosumab plus zoledronic acid at study entry, a second half-dose denosumab injection at six months, and a second zoledronic acid infusion at twelve months.

The study aims to determine whether this combined tapering-plus-bisphosphonate approach more effectively prevents lumbar spine BMD loss compared with conventional sequential therapy.

DETAILED DESCRIPTION:
Effective maintenance of bone mineral density (BMD) after discontinuing denosumab (Prolia) remains a major clinical challenge. Although denosumab is highly effective in increasing BMD, patients frequently discontinue therapy due to issues such as adherence, comorbidities, or personal circumstances. This interruption can lead to rapid and profound bone loss, substantially increasing fracture risk. Current clinical consensus recommends follow-on bisphosphonate therapy-most commonly alendronate (Fosamax) or zoledronic acid (Aclasta)-after the pharmacologic effect of denosumab wears off. However, evidence indicates that in patients treated with denosumab for more than three years, conventional bisphosphonate transition alone is often insufficient to fully prevent post-discontinuation BMD decline. Importantly, most bone loss occurs within the first year after stopping denosumab, highlighting the urgent need for strategies that can suppress the rebound increase in bone turnover during this critical period.

This study aims to investigate whether a dose-reduction (de-escalation) strategy-administering half-dose denosumab (30 mg every six months) combined with sequential zoledronic acid therapy-can better preserve lumbar spine BMD after long-term denosumab treatment. The target population includes (1) postmenopausal women with osteoporosis or osteopenia-associated fractures who have received at least three years of denosumab treatment, and (2) men aged ≥50 years with osteoporosis or osteopenia-associated fractures and ≥3 years of denosumab therapy.

The study uses an open-label, stratified randomized trial design. After enrollment, participants are stratified according to total duration of prior denosumab use: <4 years or ≥4 years. Within each stratum, participants are randomized into two groups, with 22 participants per group.

Control Group (Standard Sequential Therapy):

Participants receive conventional post-denosumab management. A single infusion of zoledronic acid is administered at the expected end of denosumab's pharmacologic effect, followed by a second zoledronic acid infusion one year later (±1 week).

Intervention Group (De-escalation + Bisphosphonate Strategy):

At study entry, participants receive a half-dose denosumab injection (expected duration of effect: six months) concurrently with one dose of zoledronic acid. Six months later (±1 week), participants receive a second half-dose denosumab injection. At twelve months after enrollment (±1 week), a second zoledronic acid infusion is administered.

This investigational regimen is designed to gradually taper denosumab exposure while simultaneously initiating bisphosphonate therapy to stabilize bone turnover. By providing partial RANKL inhibition during the early high-risk period and reinforcing mineralization with zoledronic acid, the study aims to determine whether this combined approach can more effectively mitigate the rebound effect and prevent lumbar spine BMD loss.

The results of this trial will help clarify whether a structured de-escalation plus bisphosphonate strategy offers superior protection compared with standard transition therapy in patients with long-term denosumab exposure.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged ≥50 and ≤85 years with osteoporosis- or osteopenia-related fractures who have received denosumab (Prolia) continuously for at least 3 years, with no dosing interval exceeding 9 months; and men aged ≥50 and ≤85 years with osteoporosis- or osteopenia-related fractures who have received continuous denosumab (Prolia) therapy for at least 3 years, with dosing intervals not exceeding 9 months.

Exclusion Criteria:

* Secondary osteoporosis Metabolic bone diseases Active or prior malignancy Ongoing systemic glucocorticoid therapy Current use of hormone replacement therapy Use of any medications that affect bone metabolism Estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73 m² Known hypersensitivity to zoledronic acid Hypocalcemia Any other contraindications to zoledronic acid use

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Lumbar Spine BMD Over 2 Years | 2 Years
  Change in Lumbar Spine BMD Over 2 Years

SECONDARY OUTCOMES:
Change in Total hip BMD Over 2 Years | 2 Years
  Change in Total hip BMD Over 2 Years
Change in Femoral Neck BMD Over 2 Years | 2 Years
  Change in Femoral Neck BMD Over 2 Years
Change in C-terminal telopeptide Over 2 Years | 2 Years
  Change in C-terminal telopeptide over 2 years, which reflects the level of bone resorption, will be used to assess how bone turnover responds to the intervention throughout the study period.
Change in Procollagen Type I N-Propeptide Over 2 Years | 2 Years
  Change in Procollagen Type I N-Propeptide over 2 years, which reflects the level of bone formation, will be used to assess how bone turnover responds to the intervention throughout the study period.
Incidence of clinical osteoporotic fracture | 2 years
  Incidence of clinical osteoporotic fracture

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No